CLINICAL TRIAL: NCT06135090
Title: Development and Initial Testing of a Peer-Led Trauma-Focused Intervention for Significant Others of Individuals With Borderline Personality Disorder
Brief Title: Testing a Peer-led Trauma-focused Intervention for Significant Others of Those With BPD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: York University (Other)
Collaborators: The Sashbear Foundation (Unknown)
Responsible Party: Principal Investigator, Skye Fitzpatrick, Assistant Professor, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4054
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Posttraumatic Stress Disorder; Family Members; Spouses
Keywords: Posttraumatic stress disorder; Borderline personality disorder; Peer-support; Family members; Significant others
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: The trauma recovery program (TRP) is a seven-session, peer-led, group program for family members/significant others of people with borderline personality disorder (BPD) and emotion dysregulation. It draws on principles of cognitive processing therapy for PTSD and cognitive behavioural conjoint therapy for PTSD to target PTSD symptoms in these individuals that are related to having a loved one with BPD or emotion dysregulation. As a peer-support model, it is not a psychotherapy. The TRP involves learning about common reactions to trauma and learning methods of challenging trauma-related beliefs that inhibit trauma recovery. Group members are asked to practice exercises outside of sessions that focus on challenging beliefs that fall into several key trauma-related themes.
Masking Description: This is a single arm, uncontrolled design. Thus, no masking to intervention allocation is possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma Recovery Program (official title TBD) (Experimental): The trauma recovery program (TRP) is a seven-session, peer-led, group program for family members/significant others of people with borderline personality disorder (BPD) and emotion dysregulation. It draws on principles of cognitive processing therapy for PTSD and cognitive behavioural conjoint therapy for PTSD to target PTSD symptoms in these individuals that are related to having a loved one with BPD or emotion dysregulation. As a peer-support model, it is not a psychotherapy. The TRP involves learning about common reactions to trauma and learning methods of challenging trauma-related beliefs that inhibit trauma recovery. Group members are asked to practice exercises outside of sessions that focus on challenging beliefs that fall into several key trauma-related themes.
  Interventions: Behavioral: Trauma Recovery Program (official title TBD)

INTERVENTIONS:
Behavioral: Trauma Recovery Program (official title TBD) — See arm description

SUMMARY:
This project involves developing and piloting a peer-led intervention focused on posttraumatic stress symptoms for the family members and significant others of people with borderline personality disorder. The project involves collaborating with The Sashbear Foundation who will be delivering the trauma response program (TRP) that was developed by the investigative team to its network. In phase 1 of this project, the investigators will evaluate the first delivery of the TRP at The Sashbear Foundation and solicit feedback from peer-facilitators and recipients who consent to research participation. In phase 2 of this project, the investigators will evaluate the efficacy, acceptability, and safety of the delivery of the next two to four TRPs delivered at The Sashbear Foundation consisting of up to approximately 10 group members (maximum number of TRP recipient research participants in phase 2 is 40).

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a severe mental illness characterized by intense conflict and instability in interpersonal relationships, emotion dysregulation and inappropriate anger, chronic feelings of emptiness, impulsivity, and self-injury with suicidal or non-suicidal intent. Significant others of people with BPD such as family members, friends, and intimate partners, find self-injury intensely distressing and traumatizing. Perhaps as a result, approximately two thirds of significant others of people with BPD report desiring mental health support for themselves, but not being able to access any. A recent needs assessment conducted by the investigative team involving 157 significant others of people with borderline personality disorder (BPD) suggested that 85.7% of significant others reported having traumatic experiences related to their loved one with BPD and 48.7% exhibited clinically significant posttraumatic stress disorder (PTSD) symptoms. Further, 94.8% of these individuals reported desiring an intervention focused on reducing PTSD symptoms and related phenomena. However, no interventions for significant others focused on trauma currently exist. Therefore, the investigative team collaborated to develop a peer-led, trauma-focused intervention for significant others of people with BPD and emotion dysregulation. The Sashbear Foundation is a non-profit organization that currently delivers over 1000 peer-led groups for significant others of people with BPD and related problems per year focused on education and skills to support those with BPD. The Sashbear Foundation intends to deliver the trauma response program (TRP) that was developed by the investigative team to its network, and members of the investigative team intend to provide training and consultation to members of the Sashbear Foundation regarding the delivery of TRP.

This project involves members of the investigative team providing training/consultation to members of the Sashbear Foundation, regarding the optimal delivery of TRP. It also involves an evaluation of up to the first five TRP administrations that the Sashbear Foundation is delivering. In phase 1 of this project, the investigative team will evaluate the first delivery of the TRP at The Sashbear Foundation and solicit feedback from peer-facilitators and recipients who consent to research participation. This feedback will be used to refine the TRP manual. Recipients receiving the first TRP group at The Sashbear Foundation will specifically be invited to participate in this research which involves completing measures of PTSD, other mental health and wellness outcomes, and intervention satisfaction. These measures will be administered at baseline, the half-way point, and at the end of the intervention. TRP recipients will also be invited to complete exit interviews at the end of the intervention. Feedback regarding the manual will also be informally-solicited from peer-facilitators throughout intervention delivery, leading to refinement of the intervention.

In phase 2 of this project, the investigative team will evaluate the efficacy, acceptability, and safety of the delivery of the next two to four TRPs delivered at The Sashbear Foundation consisting of up to approximately 10 group members (maximum number of TRP recipient research participants in phase 2 is 40). TRP recipients at The Sashbear Foundation who consent to participate in research procedures will complete measures of PTSD, other mental health and wellness outcomes, and intervention satisfaction. These measures will be administered at baseline, the half-way point, the end of intervention, one month after the end of intervention, and three months after the end of intervention. Phase 1 and Phase 2 TRP peer-facilitators will also be invited to complete exit interviews with the research team following the end of the intervention to capture their experiences administering TRPs.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as having experienced a trauma related to their loved one with BPD or related problems that impacts them
* Has previously received the Family Connections program at Sashbear (i.e., a peer-led intervention that teaches family members skills for managing their relationships with their loved one with BPD and related problems)

Exclusion Criteria:

* Engagement in suicidal or self-injurious behaviour in the past year
* Elevated BPD symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This 20-item measure assesses post-traumatic stress symptoms

SECONDARY OUTCOMES:
Trauma Related Guilt Inventory (TRGI) | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 32-item self- report measure that is designed to measure guilt experienced as a result of a traumatic event. It is composed of three subscales including guilt cognitions, distress, and global guilt.
Generalized Anxiety Disorder 7 (GAD-7) | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 7-item self-report scale that assesses anxiety with excellent psychometric properties.
Patient Health Questionnaire- 9 (PHQ-9) | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 9-item self-report questionnaire that assesses depression.
Burden Assessment Scale (BAS) | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 19-item self- report questionnaire that assesses burden in caregivers of individuals with a close other with serious mental illness.
Perceived Stress Scale (PSS) | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 10-item self- report questionnaire that assesses the degree to which individuals perceive life situations as stressful.
Experience of Shame Scale | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  The is a 25-item self- report questionnaire that assesses feelings of embarrassment, self- consciousness, and shame.
Brief Coping Orientation to Problems Experienced Inventory (Brief-COPE) | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  The is a 28-item self- report questionnaire that assesses coping styles in response to hardship.
Difficulties in Regulating Emotion Scale (DERS) | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 36-item self- report scale measuring emotion dysregulation.
Single items from the WHOQOL-100 | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  3 items from the 100-item self-report questionnaire will be used to measure perceived health, work functioning, and quality of life
Dyadic Adjustment Scale - 1 item | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  1 item from this self- report measure will be used to assess satisfaction with the relationship with one's close other with BPD/emotion dysregulation
Ineffective Arguing Inventory | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is an 8-item self- report measure that assesses the quality of arguments between the individual in the study and their close other with BPD/emotion dysregulation.
The Family Questionnaire | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 20-item measure that assesses expressed emotion in the context of having a close other with serious mental illness.
Posttraumatic Growth Inventory | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 21-item measure that assesses growth and self-improvement that follows a stressful encounter.
Self Compassion Scale-Short form | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 12-item self- report questionnaire that assesses one's self- compassion.
Brief Resilience Scale | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 5-item self-report measure that assesses the ability to bounce back from stressors.
Posttraumatic Cognitions Inventory-self blame subscale | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  This is a 5-item subscale that examines the extent to which people feel self- blame for traumatic experiences
PANAS-hostility scale | Baseline, 3-4 weeks, 7 weeks, 13 weeks (phase 2 only), 17 weeks (phase 2 only).
  Six items measuring past week anger/hostility.
Client Satisfaction Questionnaire | 7 weeks
  This is an 8-item scale examining the extent to which people feel satisfied with the program they received

CONTACTS AND LOCATIONS:
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data from Phase 2 will be de-identified and posted on an online and public data repository in order to promote integrity of the research and allow other researchers to replicate our findings using this data.
Supporting Information: Analytic Code